CLINICAL TRIAL: NCT02522832
Title: Discovering New Treatments for Asthma and COPD. The Use of the Human Viral Challenge Model With a Newly Manufactured and Characterised GMP Wild-Type Human Rhinovirus
Brief Title: Discovering New Treatments for Asthma and COPD. A New Human Rhinvovirus for Human Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RVL-CS-002
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Rhinovirus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Titre 1 (Experimental): Low infectious titre of innoculum
  Interventions: Other: Titre 1
- Titre 2 (Experimental): Medium infectious titre of innoculum
  Interventions: Other: Titre 2
- Titre 3 (Experimental): High infectious titre of innoculum
  Interventions: Other: Titre 3

INTERVENTIONS:
Other: Titre 1 — Virus infection
  Arms: Titre 1
Other: Titre 2 — Virus infection
  Arms: Titre 2
Other: Titre 3 — Virus infection
  Arms: Titre 3

SUMMARY:
A GMP rhinovirus was manufactured according to GMP and then characterised in human volunteers in the human viral challenge model.

DETAILED DESCRIPTION:
Human Rhinovirus infection is an important precursor to asthma and chronic obstructive pulmonary disease exacerbations and the Human Viral Challenge model may provide a powerful tool in studying these and other chronic respiratory diseases. In this study we have reported the production and human characterisation of a new HRV-16 challenge virus produced specifically for this purpose.

An HRV-16 isolate from an 18 year old experimentally infected healthy female volunteer (University of Virginia Children's Hospital, USA) was obtained with appropriate medical history and consent. We manufactured a new HRV-16 stock by minimal passage in a WI-38 cell line under Good Manufacturing Practice conditions. Having first subjected the stock to rigorous adventitious agent testing and determining the virus suitability for human use, we conducted an initial safety and pathogenicity clinical study in adult volunteers in our dedicated clinical quarantine facility in London.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults as determined by medical history, physical examination, serology (HIV and Hepatitis B and C) and clinical laboratory tests.
* Female subjects were required to provide of a history of reliable contraceptive practice.

Exclusion Criteria:included;

* asthma,
* hypersensitivity to mercurials or chicken eggs,
* anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration, chronic nasopharyngeal complaints,
* abnormal electrocardiogram (ECG),
* febrile illness or significant symptoms of upper respiratory infection on the day of
* Subjects using medication or other products for rhinitis or nasal congestion,
* Subject who had received systemic glucocorticoids within 1 month, or cytotoxic or immunosuppressive drugs within 6 months of the study start.
* Subjects agreed not to smoke during the quarantine phase.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Virus shedding defined as area under the curve | 10 days

SECONDARY OUTCOMES:
Symptoms of respiratory tract infection | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Murray, MD, Principal Investigator — PI

REFERENCES:
- [Derived] Fullen DJ, Murray B, Mori J, Catchpole A, Borley DW, Murray EJ, Balaratnam G, Gilbert A, Mann A, Hughes F, Lambkin-Williams R. A Tool for Investigating Asthma and COPD Exacerbations: A Newly Manufactured and Well Characterised GMP Wild-Type Human Rhinovirus for Use in the Human Viral Challenge Model. PLoS One. 2016 Dec 9;11(12):e0166113. doi: 10.1371/journal.pone.0166113. eCollection 2016. PMID 27936016